CLINICAL TRIAL: NCT06331559
Title: A Phase I First-in-human, Open-label Trial to Investigate the Safety, Pharmacokinetics and Antitumor Activity of SIM0501 as Monotherapy and in Combination in Participants With Advanced Solid Tumors
Brief Title: Study of SIM0501 Alone and in Combination in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company development strategy change
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Collaborators: Shanghai Xianxiang Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SIM0501-101
Record Dates: First submitted 2024-03-13; First posted 2024-03-26 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SIM0501 mono dose escalation (Experimental)
  Interventions: Drug: SIM0501 Tablets
- SIM0501 mono dose optimization (Experimental)
  Interventions: Drug: SIM0501 Tablets
- SIM0501 combination dose escalation (Experimental)
  Interventions: Drug: SIM0501 in combination with olaparib
- SIM0501 combination dose optimization (Experimental)
  Interventions: Drug: SIM0501 in combination with olaparib

INTERVENTIONS:
Drug: SIM0501 Tablets — Every 28 days is one cycle. Multiple dose levels of SIM0501 will be explored in dose escalation, and determine the maximum tolerated dose.
  Arms: SIM0501 mono dose escalation
Drug: SIM0501 Tablets — Every 28 days is one cycle.Patients will be administered a potential recommended dose of SIM0501 established from SIM0501 mono dose escalation.
  Arms: SIM0501 mono dose optimization
Drug: SIM0501 in combination with olaparib — Every 28 days is one cycle.Multiple dose levels of SIM0501 and olaparib will be explored in dose escalation, and determine the maximum tolerated dose.
  Arms: SIM0501 combination dose escalation
Drug: SIM0501 in combination with olaparib — Every 28 days is one cycle.Patients will be administered a potential recommended dose of SIM0501 combination with olaparib established from SIM0501 combination dose escalation.
  Arms: SIM0501 combination dose optimization

SUMMARY:
This is an open-label, multicenter Phase 1 clinical trial to evaluate the safety and tolerability, efficacy, and pharmacokinetics of SIM0501 in participants with advanced solid tumors. The trial consists two parts, Part 1 for SIM0501 monotherapy and Part 2 for SIM0501 in combination with olaparib. In both parts, SIM0501 with/without olaparib will be administered until disease progression or the investigator determines that continuation of the study drug would not benefit, or there is intolerable toxicity, or the participant or legal representative voluntarily requests withdrawal, or the trial is terminated.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and signature of informed consent form.
2. Aged ≥18 years, male or female.
3. Patients who have histologically confirmed advanced/metastatic solid tumors that meet the following 3 criteria: 1) progressed on at least one prior systematic anti-tumor regimen; 2) have no standard of care (SOC), or are intolerant to SOC, or have no access to SOC; 3) with documented/locally confirmed deleterious or suspected deleterious germline or somatic BRCAm, HRRm or HRD.
4. Has at least one evaluable (described below) or measurable tumor lesion according to RECIST v1.1 , and tumor lesions previously treated with radiotherapy or local therapy should be excluded as measurable lesions unless disease progression has been demonstrated. Palliative radiation therapy is allowed if there are non-radiated measurable disease in other organs.
5. Eastern Cooperative Oncology Group (ECOG) score of 0 or 1.
6. Expected survival ≥12 weeks.

Exclusion Criteria:

1. Patients unable to swallow study drug and patients with gastrointestinal disorders likely to interfere with absorption of the study drug.
2. Patient has not recovered (i.e., to Grade 1 or to baseline) from previous anticancer therapy-induced AEs.

   Note: Grade ≤2 AEs with no impact on patient safety are exceptions to this criterion and may qualify for the trial, e.g., Grade ≤2 hair loss and neuropathy caused by chemotherapy.
3. Patient is currently participating or has participated in a trial of an investigational agent or using an investigational device within 4 weeks prior to the first dose of SIM0501, including but not limited to chemotherapy, radiotherapy, target therapy, immunotherapy or other anti-cancer therapies. Note: This does not include participation in the survival follow-up of a trial.
4. Known human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS).
5. Active hepatitis B (HBsAg or HBcAb positive and HBV DNA ≥1×104 copies/mL or ≥2000 international unit [IU]/mL) or hepatitis C (HCV antibody positive and HCV RNA ≥ ULN) infection; participant with HBsAg positive or detective HBV-DNA at screening should receive antiviral treatment as per local practice during the trial.
6. Any other diseases, active or uncontrolled pulmonary dysfunction, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug, that may affect the interpretation of the results, or that renders the patient at high risk from treatment complications.
7. Patient is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2024-03-19 (Actual); Primary Completion 2025-09-17 (Actual); Study Completion 2025-09-17 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | At the end of Cycle 1 (each cycle is 28 days)
  Primary Endpoints
Adverse events will be evaluated according to the CTCAE v5.0 | The informed consent is signed until 30 days after the last dosing
  Primary Endpoints

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Cancer Hospital, Jinan, Shandong, China